CLINICAL TRIAL: NCT03490188
Title: An Innovative Patient-mentoring Program for Kidney Transplant Patients to Reduce Anxiety and Readmission Rates: a Randomized Controlled Trial Leveraging Patients
Brief Title: Design of a Standardized Patient: Mentoring Program for Kidney Transplant Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Aravind Chandrasekaran, Associate Professor, Ohio State University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017H0190
Record Dates: First submitted 2017-12-19; First posted 2018-04-06 (Actual); Last update posted 2018-08-21 (Actual); Status verified 2018-08

CONDITIONS: Kidney Transplant; Complications

STUDY DESIGN:
Intervention Model Description: A single institution randomized control trial assigning patients getting discharged after a kidney transplant to treatment and control group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Patients assigned to treatment arm will receive standard post-transplantation discharge care that includes weekly follow-up visits and 24-hour access to transplant triage call center. In addition, they will be matched with a mentor who will conduct 5 meetings with the patients (which includes one video chat meeting, 4 30-minute phone calls) and discuss the following topics related to post-discharge: Medications, Lab Work, Fluid Intake and Adherence to doctor's appointment
  Interventions: Behavioral: Discharge Mentoring
- Control Arm (No Intervention): Control arm recipient will receive standard post-transplantation discharge care that includes weekly follow-up visits and 24-hour access to transplant triage call center

INTERVENTIONS:
Behavioral: Discharge Mentoring — Phone Conversations on the importance of complying to discharge instructions delivered before discharge
  Arms: Treatment Arm

SUMMARY:
There is an increasing number in patient's undergoing kidney transplantation in the United States. Furthermore, kidney recipients have high occurrence of 30-day readmissions that leads to high hospital costs and decreased quality of life for transplant recipients. A previous research finds that high levels of post-transplant anxiety is correlated with increased likelihood of 30-day readmissions. The goal of this study is to design and implementat a randomized control trial (RCT) using a standardized post-transplant mentoring program in order to reduce 30-day readmission and post-transplant anxiety among recipients.

DETAILED DESCRIPTION:
In this research, the investigators will seek to examine the efficacy of using former patients as mentors to newly transplanted patients and its relationship with patient anxiety following discharge as well as the prevention of 30-day readmissions for kidney transplant recipients. The primary hypothesis is that the treatment group of patients who undergo a targeted mentorship program will be better compliant with the discharge instructions and will perform better when compared to the control group who undergoes current routine post-transplantation care. Evidence from this experiment can help advance our understanding of patient-engagement in the continuity of care delivery, decrease patient readmission rates, and improve overall cost utilization.

Methods:

The investigators will conduct a single institution randomized control trial assigning patients getting discharged after a kidney transplant to a treatment group that involves a 30-day mentoring initiative by former transplant patients, and comparing the efficacy with a similar control group. The overall study period will be divided into the following sections, summarized in Figure 1.

ELIGIBILITY:
Inclusion Criteria:

* any patient who received a kidney transplantation, deceased or living donor, during the study period.

Exclusion Criteria:

* anyone younger than 18 years old or older than 70 years old.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2018-11 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
30-day readmissions | 30-days

SECONDARY OUTCOMES:
Post Transplant Anxiety | 1 Day of Discharge and 30-days after discharge
  State-Trait Anxiety Inventory (STAI) for Adults
Preventable Re-admissions | 30-days after day of discharge
  Re admissions due to missed labs or medications as measured by time of readmission for any readmission that was deemed preventable by physiologic laboratory data, reason for readmission, and primary complaint determined by trained kidney transplantation nurses

CONTACTS AND LOCATIONS:
Locations (1):
- Comprehensive Transplant Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chandrasekaran A, Anand G, Sharma L, Pesavanto T, Hauenstein ML, Nguyen M, Gadkari M, Moffatt-Bruce S. Role of in-hospital care quality in reducing anxiety and readmissions of kidney transplant recipients. J Surg Res. 2016 Sep;205(1):252-259.e1. doi: 10.1016/j.jss.2016.05.032. Epub 2016 May 27. PMID 27329569